CLINICAL TRIAL: NCT03349359
Title: Impact of Cytomegalovirus (CMV) Status Prior Antiretroviral Therapy on HIV Viral Load Decay
Brief Title: Impact of CMV Status on HIV Viral Load Decay
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_006
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: HIV antiretroviral therapy — HIV patients are receiving an antiretroviral therapy according to the physician's discretion and the availability of drugs

SUMMARY:
Background: Cytomegalovirus (CMV) infection is usually observed among patients with HIV infection. No study to date has investigated the impact of CMV infection on HIV viral load decay during antiretroviral therapy.

Methods: 345 consecutive HIV patients coinfected (N=300) or not (N=45) with CMV were enrolled. Clinical, biological and virological data were collected from HIV antiretroviral therapy initiation to the day of HIV viral load undetectability if any.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients starting an antiretroviral therapy
* CMV serology available at antiretroviral therapy initiation
* HIV viral load assessed at each follow-up visit after treatment initiation

Exclusion Criteria:

* HIV antiretroviral treatment initiation before June 2005

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients followed at the Department of Infectious Diseases, Croix-Rousse Hospital, Groupement Hospitalier Nord, Hospices Civils de Lyon, Lyon, France between June 2005 and July 2016 starting an antiretroviral treatment and with available CMV serology at treatment initiation.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
HIV viral load undetectability | From date of HIV therapy initiation until the date of HIV viral load undetectability (12 weeks in average after treatment initiation)
  HIV viral load was assessed during the follow-up visits after the initiation of antiretroviral therapy. HIV undetectability was defined by an HIV-RNA level <50 copies/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No